CLINICAL TRIAL: NCT01673724
Title: Effect of Pramipexole and Bromocriptine on Nonmotor Symptoms of Early Parkinson's Disease: Multicenter, Open-label, Parallel, Randomized Study
Brief Title: Pramipexole and Bromocriptine on Nonmotor Symptoms of Early Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKL001
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole; Bromocriptine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pramipexole (Experimental): dosage form: tablet dosage: pramipexole 0.125/0.25/0.5/1mg frequency: tid duration: 24weeks
  Interventions: Drug: pramipexole
- Bromocriptine (Active Comparator): bromocriptine dosage form: white round tablet
  Interventions: Drug: Bromocriptine

INTERVENTIONS:
Drug: pramipexole — pramipexole
  Other Names: Sandoz Pramipexole
  Arms: pramipexole
Drug: Bromocriptine — bromocriptine
  Other Names: Parlodel tab
  Arms: Bromocriptine

SUMMARY:
The purpose of this study is to determine whether pramipexole and bromocriptine are effective in the treatment of non-motor symptoms in Parkinson's Disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE Evaluate the Improvement of Nonmotor symptom scale (NMSS) between Pramipexole and Bromocriptine for early Parkinson's disease during 24-week treatment

SECONDARY OBJECTIVE

* Evaluate the improvement for Depression which is one of the Nonmotor symptoms
* Evaluate the improvement of clinical symptoms between two groups
* Evaluate the improvement of Quality of Life between two groups

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease patients in accordance with UK Queensquare Brain Bank
* modified Hoehn & Yahr stage <3
* Dopamine agents(Levodopa, dopamine agonists) naive patients, or the patients who have discontinued the agents at least four weeks before the screening in case of using the dopamine agents are administered before.

Exclusion Criteria:

* K-MMSE<24
* History of drug-induced Parkinsonism
* secondary parkinsonism
* History of schizophrenia or hallucination
* Requirement of treatment with anti-depressants due to depressive disorder
* Pregnant and/or breeding women
* Renal inadequacy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-02; Primary Completion 2016-05-23 (Actual); Study Completion 2016-05-23 (Actual)

PRIMARY OUTCOMES:
K-NMSS | 24 weeks
  Evaluate The total and each category score of K-NMSS

SECONDARY OUTCOMES:
K-MADRS | 24 weeks
  Evaluate the Improvement of the depression refering to the total score of K-MADRS
UPDRS I/II/III | 24 weeks
  Evaluate the improvement of UPDRS I/II/III
K-PDQ39 | 24 weeks
  Evaluate the improvement of Patient's QOL

CONTACTS AND LOCATIONS:
Overall Officials: Seongbeom Koh, MD, Principal Investigator — Korea University Guro Hospital
Locations (7):
- South Korea (7):
  - Korea University Ansan Hospital, Ansan
  - Inje University Busan Paik Hospital, Busan
  - Youngnam University Hospital, Daegu
  - Kangwon Nat'l University Hospital, Kangwon
  - Inje university Sanggye Paik Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul